CLINICAL TRIAL: NCT03106558
Title: Post-Market Study of Robotic-Arm Assisted Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017WHoz
Record Dates: First submitted 2017-02-07; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Manual instrument total knee replacement (Active Comparator)
  Interventions: Device: Total Knee Arthroplasty using Manual Instrumentation
- Robitic arm total knee replacement (Active Comparator)
  Interventions: Device: Total Knee Arthroplasty using Robotic Arm

INTERVENTIONS:
Device: Total Knee Arthroplasty using Manual Instrumentation
  Arms: Manual instrument total knee replacement
Device: Total Knee Arthroplasty using Robotic Arm
  Arms: Robitic arm total knee replacement

SUMMARY:
This is an early user evaluation of the robotic-assisted total knee arthroplasty platform. The objective of this surgeon group is to capture data on the defined objectives and provide Stryker with feedback.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires primary total knee surgery
* Patient is willing and able to comply with postoperative follow-up requirements and self evaluations
* Patient is willing to sign an IRB approved informed consent
* Patient is at least 18 years of age

Exclusion Criteria:

* Patient has a BMI > 50
* Patient is skeletally immature
* Patient has an active infection or suspected infection in or about the joint
* Bone stock that is inadequate to support fixation of the prosthesis
* Neuromuscular disorders, muscular atrophy or vascular deficiency in the affected limb rendering the procedure unjustified.
* Patients with mental or neurological conditions which may be incapable of following instructions.
* Blood supply limitations
* Collateral ligament insufficiency.
* Patients with prior HTOs or Unis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Component alignment | 6 weeks post knee arthroplasty
  CT scan measurement

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Athens Orthopedic Clinic, Athens, Georgia
  - Rothman Institute, Egg Harbor, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Rothman Institute, Philadelphia, Pennsylvania